CLINICAL TRIAL: NCT03390153
Title: Reduction of Shear Forces Using Semi-flexible Sockets on Transtibial Amputees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Gurinder Bains, Associate Professor, Loma Linda University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 5170454
Record Dates: First submitted 2017-12-14; First posted 2018-01-04 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Amputation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- semi flexible socket group (Experimental): A new form of residuum containment is the semi-flexible carbon fiber prosthetic socket. A semi-flexible carbon fiber socket is constructed with the same security for the subject in mind, and is even more lightweight than a rigid socket. The carbon fiber and resin used in a semi-flexible socket may provide the same durability and stability as previous designs, but will deform, intentionally, without failing (breaking). This distinct feature of semi-flexible sockets makes them a potential option for people living with limb loss. By moving slightly with the residual limb, the socket-user-interface should experience fewer forces/stresses, and yield greater comfort for the prosthetic user.
  Interventions: Other: semi flexible socket
- rigid fiber socket group (Active Comparator): A rigid carbon fiber socket is constructed for security and is mechanically lightweight to ensure stability and efficient build height. Carbon is used for its durability and stability. It proves to be a detriment in comfort and flexibility. The standard for carbon fiber weaves come in two forms: Unidirectional (UD) and Bidirectional (BD). UD carbon fiber has a zero-degree alignment, which is highly durable when compressed, but has low torsional durability. The BD carbon fibers are aligned in a 90 degree angle allowing for moderate compression and torsional strength. When oriented at 45 degrees to the line of progression, fibers become more flexible and exhibit greater torsional strength. Resins and glass composites are added to ensure security and sturdiness.
  Interventions: Other: rigid fiber socket

INTERVENTIONS:
Other: semi flexible socket — The investigators will analyze the subject's gait by trained visual diagnosis and video gait analysis, to determine comfort and safety. Any modifications will be done at this time. Once the subjects, student, and faculty investigators are satisfied with the overall fit of prostheses, a student investigator will insert force sensors into the socket to evaluate pressure. In the 'Comfort Test', walk at a self-selected pace on a treadmill for 10 minutes. Subjects will then perform a single stance activity on a Balance Master. Investigators will remove the force sensors and do one final safety check of prostheses before each subject takes their definitive socket home. Subjects will be required to wear the prosthesis given to them for one week before returning for a follow up appointment.
  Arms: semi flexible socket group
Other: rigid fiber socket — The investigators will analyze the subject's gait by trained visual diagnosis and video gait analysis, to determine comfort and safety. Any modifications will be done at this time. Once the subjects, student, and faculty investigators are satisfied with the overall fit of prostheses, a student investigator will insert force sensors into the socket to evaluate pressure. In the 'Comfort Test', walk at a self-selected pace on a treadmill for 10 minutes. Subjects will then perform a single stance activity on a Balance Master. Investigators will remove the force sensors and do one final safety check of prostheses before each subject takes their definitive socket home. Subjects will be required to wear the prosthesis given to them for one week before returning for a follow up appointment.
  Arms: rigid fiber socket group

SUMMARY:
The purpose of this graduate student research study, is to test two different sockets for comfort and test what pressures are created by the socket during daily activities. The objective is to illustrate that semi-flexible sockets will maintain its rigidity and resist progressive shear forces from daily activity, ergo making our prosthetic system a more comfortable experience for the prosthetic user.

DETAILED DESCRIPTION:
Subjects will immediately be prepared for a casting of their residual limb. On the second visit, subjects will return to be fitted with a definitive rigid carbon fiber socket. At this time, a questionnaire and physical assessments will determine subjects comfort and safety. The physical assessment consists of a ten minute walk on a treadmill, at a self-selected pace. A balancing test on a SMART Balance Master will also be used to assess subject safety, by utilizing the limits of stability protocol. Subjects' will be required to wear the prosthesis given to them for one week before returning for a follow-up appointment. On the third visit, the subjects' will return the first prosthesis to the investigators of the study, where an additional socket will be given to the subject for the second portion of this study. Subjects will be evaluated with a questionnaire and physical assessments to determine comfort and safety. Participants will be required to wear the prosthesis given to them for one week before returning for a follow-up appointment. During the final appointment, the subjects will return all devices given to them to an investigator of the study.

ELIGIBILITY:
Inclusion Criteria:

* Transtibial amputee with mature limb
* Minimum of 3-years of prosthetic use
* Capable of ambulating on a treadmill for ten minutes
* Minimum age of 18 years old
* Both Unilateral and Bilateral Amputees
* K-Level K2-K4

Exclusion Criteria:

* Any open wounds/ulcerations on the residual limb
* Skin allergies to silicone or latex
* Unmanaged co-morbidities such a diabetes and congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Balance | Change in balance between Week 2 and Week 3 of study
  The SMART Balance Master is a device used to measure balance. It consists of a plate with force sensors that can measure the subject's center of gravity as the subject shifts their position back and forth through the exercise. We will be exerting the subjects through the different phases of gait also known as a Limits of Stability test, one of the many pre-programed tests available to choose from.The SMART Balance Master is a widely used device in the rehabilitation world to test an individual's balance and ascertain their functional limits. It is a device that has great repeatability and is used to test individuals rehabilitation progress. It is also used extensively in research due to its high reproducibility. The SMART Balance Master is manufactured by Natus Medical Incorporated which is located in Pleasanton California.

SECONDARY OUTCOMES:
Socket liner integrity | Change in socket liner between Week 2 and Week 3 of study
  The Socket Liner Integrity Checklist (SLIC) has been developed by one of our student investigators which has worked in the industry for 9 years. The SLIC will be used to evaluate the wear that the socket exerts on the liner. We hypothesize that semi-flexible sockets will reduce wear of the liner, and we will use the SLIC to evaluate. The semi-flexible socket will also need to be evaluated. A semi-flexible socket might be a more comfortable experience for the user but if it does not hold up to the rigours of daily activities wear and tear, it is not a better alternative. This checklist will focus on specific areas of that socket which are prone to failure to more easily catch any major flaws.

CONTACTS AND LOCATIONS:
Overall Officials: Gurinder Bains, PhD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda Universtiy, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No